CLINICAL TRIAL: NCT03925883
Title: Predicting and Addressing Colonoscopy in Safety Net Settings
Acronym: PRECISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Sea Mar Community Health Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 1R01CA218923-01A1 (NIH); R01CA218923 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2022-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; Cancer screening; Risk prediction model; Patient navigation; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Navigation (Active Comparator): Patients randomized to this arm will receive patient navigation with the goal of completing a follow-up colonoscopy within 12 months of a positive FIT result.
  Interventions: Behavioral: Patient navigation
- Usual Care (No Intervention): Patients will receive usual care screening opportunities

INTERVENTIONS:
Behavioral: Patient navigation — Receive up to 6 live phone calls with a patient navigator for education, barrier assessment, and barrier resolution to follow up colonoscopy
  Arms: Patient Navigation

SUMMARY:
The prospective cohort study will evaluate the effectiveness of patient navigation in community health center settings. The investigators will collaborate with the advisory board, composed of key clinicians and patients, researchers, and policymakers, to establish a procedure to conduct and evaluate a patient navigation program that aims to increase rates of follow-up colonoscopy among diverse patient populations served by safety net clinics. Phase 1 will be a milestone-driven planning process in which the investigators will validate the risk prediction model and apply the risk prediction model to stratify the patients and adapt patient navigation materials for the local context. Phase II will be a large-scale, patient randomized-controlled trial that will include 1200 patients at a large 34-clinic community health center in Washington State.

DETAILED DESCRIPTION:
The study will fulfill the following aims:

Aim 1: Validate externally the predictive risk score using Sea Mar CHC's robust data including 29,000 patients age-eligible for colorectal cancer screening; stratify patients according to risk of non-adherence to follow-up colonoscopy; and adapt patient navigation program for the local context.

Aim 2: Assess the effectiveness, costs, and cost-effectiveness of a centralized, phone-based patient navigation program for follow-up colonoscopy receipt for patients at moderate risk or high risk for non-adherence.

Aim 3: Assess differences in the intervention arms in secondary outcomes (e.g. time to colonoscopy receipt, no-show/canceled appointments, colonoscopy quality) and moderators of intervention effectiveness (e.g. probability level, intervention dose, and patient age, ethnicity, and sex)

ELIGIBILITY:
Inclusion Criteria:

* Positive FIT test

Exclusion Criteria:

* Prior colorectal cancer
* Dialysis patient

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-06-05 (Actual); Study Completion 2023-06-05 (Actual)

PRIMARY OUTCOMES:
Rate of follow-up colonoscopy | 12 months
  Receipt of colonoscopy within 1 year of abnormal Fecal Immunochemical Test (FIT) result

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Coronado, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States

REFERENCES:
- [Derived] Coronado GD, Petrik AF, Thompson JH, Leo MC, Slaughter M, Gautom P, Hussain SA, Mosso L, Gibbs J, Yadav N, Mummadi RR, Johnson ES, Jimenez R. Patient Navigation to Improve Colonoscopy Completion After an Abnormal Stool Test Result : A Randomized Controlled Trial. Ann Intern Med. 2025 May;178(5):645-654. doi: 10.7326/ANNALS-24-01885. Epub 2025 Apr 1. PMID 40163863
- [Derived] Coronado GD, Kihn-Stang A, Slaughter MT, Petrik AF, Thompson JH, Rivelli JS, Jimenez R, Gibbs J, Yadav N, Mummadi RR. Follow-up colonoscopy after an abnormal stool-based colorectal cancer screening result: analysis of steps in the colonoscopy completion process. BMC Gastroenterol. 2021 Sep 28;21(1):356. doi: 10.1186/s12876-021-01923-1. PMID 34583638
- [Derived] Coronado GD, Johnson ES, Leo MC, Schneider JL, Smith D, Mummadi R, Petrik AF, Thompson JH, Jimenez R. Patient randomized trial of a targeted navigation program to improve rates of follow-up colonoscopy in community health centers. Contemp Clin Trials. 2020 Feb;89:105920. doi: 10.1016/j.cct.2019.105920. Epub 2019 Dec 24. PMID 31881390

DOCUMENTS (2):
  • Study Protocol (2022-12-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03925883/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT03925883/SAP_001.pdf